CLINICAL TRIAL: NCT02331693
Title: Genetically Modified T Cells in Treating Patients With Malignant Gliomas Overexpressing EGFR
Brief Title: CAR T Cells in Treating Patients With Malignant Gliomas Overexpressing EGFR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-20141110
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Glioma
Keywords: EGFR; CAR T cells; glioma
MeSH Terms: conditions — Glioma

ARMS (1):
- anti-EGFR CAR T (Experimental)
  Interventions: Biological: anti-EGFR CAR T

INTERVENTIONS:
Biological: anti-EGFR CAR T
  Other Names: CAR T cells targeting overexpressed EGFR in cancer cells

SUMMARY:
The purpose of this study is to determine whether autologous T cells bearing chimeric antigen receptor that can specifically recognize EGFR overexpressed in tumor cells is safe and effective for patients with EGFR-overexpressing malignant glioma.

DETAILED DESCRIPTION:
BACKGROUND:

- Patients with advanced gliomas have very limited treatment options. Epidermal Growth Factor Receptor (EGFR) is often amplified in patients with glioblastoma (GBM) and has been regarded a suitable target for GBM treatment.

The investigators have constructed lentiviral vector that contains a chimeric antigen receptor (CAR) that recognizes overexpressed EGFR in tumor cells but not EGFR in normal cells, which can be used to mediate genetic transfer of this CAR with high efficiency without the need to perform any selection.

OBJECTIVES:

Primary Objectives To evaluate the safety of the administration of anti-EGFR CAR engineered T lymphocytes in patients receiving the non-myeloablative conditioning regimen, and aldesleukin

Secondary objectives To determine whether the glioma will regress after the patients receive anti-EGFR CAR-engineered T lymphocytes and aldesleukin following a nonmyeloablative but lymphoid depleting preparative regimen.

ELIGIBILITY:

Histologically proven glioblastoma or glisarcoma overexpressing EGFR as determined by IHC, Western blot, FISH or RT-PCR.

Failed prior standard treatment with radiotherapy with or without chemotherapy. Cardiac, pulmonary and laboratory parameters within acceptable limits

DESIGN:

The study will be conducted using a Phase I design. Patients will receive a non-myeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumor reactive, CAR gene-transduced T cells, plus IV aldesleukin.

A total of 10 patients may be enrolled over a period of 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven glioblastomas or gliosarcomas that overexpress EGFR as assessed by IHC, FISH, western blot or RT-PCR.
2. Patients must have progression of disease after radiotherapy (including patients that undergo surgery for recurrent disease and are rendered NED). This includes recurrent GBM after receiving all standard first-line treatment, including surgery (if feasible due to neurosurgical and neuro-anatomical considerations) and adjuvant radiotherapy +/- chemotherapy.
3. Patients must either not be receiving steroids, or be on a stable dose of steroids for at least five days prior to registration.
4. Patients must be greater than or equal to 18 years of age and less than or equal to age 70, and must have a life expectancy > 8 weeks
5. Patients must be able to understand and sign the Informed Consent Document
6. Must be willing to sign a durable power of attorney.
7. Patients of both genders must be willing to practice birth control for four months following treatment.
8. Women of child bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
9. Serology:

   Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.) Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
10. Hematology WBC greater than or equal to 3000/mm(3) ANC greater than or equal to 1000/mm(3) without the support of filgrastim Platelet count greater than or equal to 100,000/mm(3) Hemoglobin greater than or equal to 8.0 g/dl (eligibility level for hemoglobin may be reached by transfusion)
11. Chemistry:

    ALT/AST less than or equal to to 2.5 times the upper limit of normal Creatinine less than or equal to to 1.6 mg/dl Total bilirubin less than or equal to to 1.5 mg/dl, except in patients with Gilbert s Syndrome who must have a total bilirubin less than 3.0 mg/dl.
12. Patients must be at least 4 weeks from radiation therapy. Additionally, patients must be at least 6 weeks from nitrosoureas, 4 weeks from temozolomide, 3 weeks from procarbazine, 2 weeks from vincristine and 4 weeks from last bevacizumab administration. Patients must be at least 4 weeks from other cytotoxic therapies not listed above and 2 weeks for non-cytotoxic agents (e.g., interferon, tamoxifen) including investigative agents. All toxicities from prior therapies should be resolved to CTCAE less than or equal to grade 1 (except for toxicities such as alopecia, or vitiligo).

Exclusion Criteria:

1. A prior history of gliadel implantation in the past six months..
2. Women who are currently pregnant or breast feeding because of the potentially dangerous effects of the treatment on the fetus or infant.
3. Active systemic infections, coagulation disorders or other major medical illnesses including those of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
6. History of severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, or aldesleukin.
7. History of coronary revascularization or ischemic symptoms.
8. Clinically significant hemorrhagic or ischemic stroke, including transient ischemic attacks and other central nervous system bleeding in the preceding 6 months that were not related to glioma surgery. History of prior intratumoral bleeding is not an exclusion criteria; patients who with history of prior intratumoral bleeding, however, need to undergo a non-contrast head CT to exclude acute bleeding.
9. Other concomitant anti-cancer therapy except corticosteroids.
10. Any patient known to have an LVEF less than or equal to 45%.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events attributed to the administration of the anti-EGFR CAR T cells | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Institute, Xuhui, Shanghai Municipality, China